CLINICAL TRIAL: NCT07215286
Title: Comparative Study on SNAG From Loaded and Unloaded Position in the Treatment of Low Back Pain
Brief Title: Comparative Study on SNAG From Different Positions Low Back Pain Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Kamel Ahmed, Assistant Professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2025-910
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Non Specific Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loaded-SNAG (Active Comparator): SNAGs from standing position
  Interventions: Procedure: Loaded-SNAG; Procedure: Unloaded-SNAG
- Unloaded-SNAG (Active Comparator): SNAG from quadruped position
  Interventions: Procedure: Loaded-SNAG; Procedure: Unloaded-SNAG

INTERVENTIONS:
Procedure: Loaded-SNAG — patients will receive SNAGs from standing (Loaded-SNAG), step-stance, or functional position that provokes symptoms. A specialized Mulligan belt was used around the patient's waist and the therapist's hips. The mobilizing force was applied parallel to the facet joint plane (cephalic direction) and over the spinous processes of the respective symptomatic spinal levels. The therapist's hand's ulnar aspect was used over the spinous process of the superior vertebra of the involved segment for flexion glide. The therapist applies accessory glide to targeted zygapophyseal level while the patient actively performs symptomatic movement (e.g., forward flexion), performing repetitions with the therapist maintaining the glide.
Procedure: Unloaded-SNAG — patients will receive unloaded SNAG from quadruped position to reduce the axial loading. The therapist applies the equivalent accessory glide at the symptomatic spinal level while the patient performs the symptomatic movement (modified to be non-weight-bearing).

SUMMARY:
Background: Low back pain (LBP) is a leading cause of disability worldwide. Mulligan's Sustained Natural Apophyseal Glides (SNAGs) are manual therapy techniques shown to reduce pain and improve function in LBP. However, whether applying SNAGs in loaded (weight-bearing) versus unloaded (non-weight-bearing) positions yields superior clinical outcomes remains unclear.

Objective: To compare the effects of lumbar SNAGs applied in loaded versus unloaded positions on pain, disability, and function in individuals with chronic non-specific LBP.

Methods: A randomized, single-blind, parallel-group clinical trial will recruit 34 participants with chronic LBP. Participants will be allocated to receive SNAGs in either loaded or unloaded positions, combined with a standardized exercise program, for 6 sessions over 1 week. The primary outcome is pain intensity (Numeric Pain Rating Scale) and lumbar flexion range of motion. Secondary outcomes include disability (Oswestry Disability Index). Outcomes will be measured at baseline and immediately post-treatment. Data will be analyzed using linear mixed models on an intention-to-treat basis.

Conclusion: This trial will determine whether a loaded SNAG application provides superior benefits compared to unloaded SNAG in the treatment of chronic LBP. Findings may guide clinical decision-making and optimize manual therapy application.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non specific low back pain for 6 weeks or more
* Who scored between three and six on a visual analogue scale (VAS)
* Restriction of the movement was only in flexion ROM

Exclusion Criteria:

* Pregnancy,
* Obese,
* Infectious conditions of the spine,
* Autoimmune disorders,
* Malignancy
* Any contraindication to physiotherapy and manual therapy
* Any patient received physical therapy sessions last 6 months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 1 week
  Visual analogue scale (VAS), which is a 10-cm line, 0 denotes no pain and 10 the most intense agony.
Lumbar flexion ROM | 1 week
  The BROM is an electronic goniometer that will be used to evaluate the range of motion for trunk flexion

SECONDARY OUTCOMES:
Functional disability | 1 week
  The functional level was assessed using a validated Arabic version of the Oswestry Disability Index (ODI). A total score will be calculated, the percentage of disability (score obtained divided by 50 and multiplied by 100) ranged from 0% (no disability) to 100% (complete disability).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Clinics, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The project is funded by university of Hail and all the data should be authorized through it